CLINICAL TRIAL: NCT05927545
Title: The Efficacy of Manual Therapy and BETY on Headache and Quality of Life in Patients With Temporomandibular Dysfunction Related Headache
Brief Title: Efficacy of Manuel Therapy and BETY in Patients With Temporomandibular Dysfunction Related Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Feride ATAY, PT, Msc, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-101
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2024-08

CONDITIONS: Temporomandibular Disorders; Headache
Keywords: Temporomandibular Disorders, Headache, Quality of Life, Pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Headache; Pain | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home Exercise: Patient Education and Preventive Exercise (Active Comparator): Group 1: The home Exercise Program includes an educational training program about parafunctional activities and correction exercises for patients having TMD-related headaches. The program includes tongue resting position, diaphragmatic breathing, head posture correction exercises, stretching and strengthening exercises for shoulder and back muscles, and active cervical and thoracic mobilization.
  Interventions: Procedure: Patient education and preventive exercise
- Manual Therapy Combined with Home Exercise (Active Comparator): Group 2: MT group includes in addition to the home exercise program, deep friction massage, myofascial release techniques and stretching techniques to masticatory and neck muscles, temporomandibular joint and cervical mobilization will be applied.
  Interventions: Procedure: Patient education, preventive exercise combined with Manual Therapy protocol
- Cognitive Exercise Therapy Approach Combined with Home Exercise (Active Comparator): Group 3: Cognitive Exercise Therapy Approach (CETA) includes cognitive exercise therapy and the home exercise program. The Cognitive Exercise Therapy approach is an innovative exercise approach that aims to change the patient's cognition about the disease through exercise and is suitable for the biopsychosocial model. CETA is an exercise approach aimed at changing the patient's cognitive perception of the disease through exercise, placing the responsibility of disease management on the patient. The approach will be explained in the first session, and patients will be taught proper posture for the neck, shoulders, thoracic, and lumbopelvic region, as well as correct breathing control. Each 1-hour session will include a warm-up, exercise period, and cool-down.
  Interventions: Procedure: Patient education, preventive exercise combined with BETY approach

INTERVENTIONS:
Procedure: Patient education and preventive exercise — Educational training program and prevention exercises about temporomandibular dysfunction in patients with temporomandibular dysfunction-associated headaches.
  Arms: Home Exercise: Patient Education and Preventive Exercise
Procedure: Patient education, preventive exercise combined with Manual Therapy protocol — Manual therapy program combined with the educational training program and prevention exercise about temporomandibular dysfunction in patients with temporomandibular dysfunction-associated headaches.
  Arms: Manual Therapy Combined with Home Exercise
Procedure: Patient education, preventive exercise combined with BETY approach — BETY therapy program combined with the educational training program and prevention exercise about temporomandibular dysfunction in patients with temporomandibular dysfunction-associated headaches.
  Arms: Cognitive Exercise Therapy Approach Combined with Home Exercise

SUMMARY:
The aim of the study is to investigate the effects of Manual Therapy and the Cognitive Exercise Therapy Approach treatment in patients with TMD-related headaches.

DETAILED DESCRIPTION:
60 subjects with TMD-related headaches, according to ICHD-3, will be included in the study after the voluntary consent form will be filled out. Subjects will randomly be divided into 3 groups according to the order.

Group 1: Patient education and exercise group: The patients in this group will be taught an exercise program after general education. Education training program about parafunctional activities of TMD and active exercises for masticatory and neck muscles. Patients will be asked to complete and follow-up home exercises for 30-45 minutes once a day, 5 days a week for 8 weeks. The continuity of the exercises will be ensured by sending reminder messages to this group of patients about doing their exercises once a week by the physiotherapist.

Group 2; Manuel Therapy group: This group will receive the same patient education and exercises additionally manual therapy program which is planned to last 45 minutes will be applied twice a week, for 8 weeks.

Group 3; BETY group: This group will receive the same patient education and exercises in addition BETY approach, which is the Cognitive Exercise Therapy Approach treatment, will be applied in 2 sessions a week for 45 minutes and a total of 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 60 years old
* Getting a diagnosis of TMD-related headache
* Not having received FTR and manual therapy in the last 3 months
* Having pain ≥ 50 or more according to the headache impact test (HIT 6)
* Patients who have not received medical treatment in the last 3 months and will not receive medical treatment during the treatment
* Patients who describe pain in the jaw, face, temporal region or ear for at least 6 months and who have pain in the chewing muscles with palpation

Exclusion Criteria:

* Ages under 18 and over 60 years old
* Patients with disc displacement and/or attachment degeneration
* Patients with dental infection
* Patients who have undergone facial and ear surgery in the last six months
* Patients undergoing orthodontic treatment
* Patients using regular analgesics or anti-inflammatory drugs
* Patients with a history of trauma (whiplash injury, condylar trauma, fracture),
* Patients who have undergone any surgery related to the cervical and/or TMJ
* Patients with facial paralysis
* Patients with missing teeth in the upper jaw
* Patients with cognitive deficits
* Participation rate lower than 80% of the program schedule

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-05-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Pain at 8 weeks and 5 months | Baseline, 8 weeks, 5 months
  A visual Analog Scale will be used where patients will be asked to rate their pain on a scale from 0 to 10 with 0 indicating no pain and 10 the maximum worst pain, at the baseline and the end of 8 weeks of intervention and at the end of 5 months from baseline.
Change from baseline in McGill Pain Questionnaire (SF-MPQ) at 8 weeks and 5 months | Baseline, 8 weeks, 5 months
  A short form of the McGill Pain Questionnaire (SF-MPQ) will be used. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors.
Change from baseline in pain threshold at 8 weeks and 5 months | Baseline, 8 weeks, 5 months
  A digital pressure pain threshold algometer measuring device will be used to narrow trigger point sensitivity (Wagner Instruments, Greenwich, USA). Pain measurements of pressure to the masseter, temporal, SCM, upper trapezius, suboccipital, and levator scapula muscles will be recorded.
Change from baseline in the Headache Impact Test (HIT-6) at 8 weeks and 5 months | Baseline, 8 weeks, 5 months
  The HIT-6 consists of six items: pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress. The patient answers each of the six related questions using one of the following five responses: "never", "rarely", "sometimes", "very often", or "always". These responses are summed to produce a total HIT-6 score that ranges from 36 to 78, where a higher score indicates a greater impact of headache on the daily life of the respondent. Scores can be interpreted using four groupings that indicate the severity of headache impact on the patient's life.
Change from baseline head posture analysis at 8 weeks and 5 months | Baseline, 8 weeks, 5 months
  Head posture will be measured in degrees with the goniometer as the angle between the horizontal plane and the seventh cervical vertebra and the ear line.
Change from baseline in the evaluation of Temporomandibular Joint (TMJ) and Cervical Region Range of Motion (ROM) at 8 weeks and 5 months | Baseline, 8 weeks, 5 months
  TMJ ROM: A linear ruler will be used for maximal mouth opening, right and left lateralization, and protrusion values by looking at active and passive.
  Cervical ROM: In order to measure its patency, the cervical region flexion, extension, right-left lateral flexion, and right-left rotation degrees will be measured and recorded with a goniometer.
Change from baseline in the viscoelastic properties at 8 weeks and 5 months | Baseline, 8 weeks, 5 months
  A digital MyotonPro (Myoton AS, Estonia) instrument measuring device will be used to evaluate the viscoelastic properties of the facial and neck muscles.
Change from baseline in jaw function limitation at 8 weeks and 5 months | Baseline, 8 weeks, 5 months
  Jaw function limitation will be measured by the Jaw Functional Limitation Scale-20 (JFLS-20) where the patients will be asked from 1 to 10 points per item (higher scores indicate worse jaw function). The JFLS-20 has 3 subscales: Mastication (6 items), Vertical Jaw Mobility (4 items), and Emotional and Verbal Expression (10 items).
Change from baseline in the neck disability index at 8 weeks and 5 months | Baseline, 8 weeks, 5 months
  The neck disability index (NDI) has become a standard tool for measuring self-assessed disability due to neck pain. Each of the 10 items receives a score from 0 to 5. The maximum score is 50.Scoring intervals for interpretation; 0 to 4 = no disability, 5 to 14 = mild, 15 to 24 = moderate, 25 to 34 = severe, Above 34 = complete
Change from baseline in the Pittsburgh sleep quality index at 8 weeks and 5 months | Baseline, 8 weeks, 5 months
  The Pittsburgh Sleep Quality Index (PUKI) will be used to assess sleep quality. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Change from baseline in Fatigue severity at 8 weeks and 5 months | Baseline, 8 weeks, 5 months
  The fatigue severity scale has nine items. For each question, the patient is asked to choose a number from 1 to 7 that indicates how much the patient agrees with each statement, where 1 indicates strong disagreement and 7 indicates strong agreement. A score of 4 or higher generally indicates severe fatigue.
Change from baseline in anxiety and depression at 8 weeks and 5 months | Baseline, 8 weeks, 5 months
  Hospital Anxiety and Depression scale consists of 14 questions in total. The minimum score for the anxiety and depression subscales is 0, and the maximum score is 21. An increase in the score on the scale means that the severity of anxiety and depression increases. The cut-off points were determined as 10 for the anxiety subscale and 7 for the depression subscale.
Change from baseline in Quality of Life-Oral health impact profile-14 at 8 weeks and 5 months | Baseline, 8 weeks, 5 months
  The quality of life will be evaluated with Quality of Life-Oral health impact profile-14 (OHIP-14) questionnaire. The index provides a comprehensive measure of self-reported dysfunction, discomfort, and disability resulting from oral conditions whose dimensions are based on Locker's conceptual model of oral health. Responses are rated on a 5-point Likert scale: 0 = never; 1 = hardly ever; 2 = occasionally; 3 = quite often; 4 = very often/every day. OHIP-14 scores can range from 0 to 56 and are calculated by adding the rank values for 14 items. Area scores can range from 0 to 8. Higher OHIP-14 scores indicate worse, lower scores indicate better OHRQol.
Change from baseline in Cognitive Exercise Therapy Approach Questionnaire at 8 weeks and 5 months | Baseline, 8 weeks, 5 months
  It is a measurement tool developed in accordance with the biopsychosocial model and evaluating the biopsychosocial status of patients with rheumatic disease. This scale consists of 30 items and consists of questions assessing cognitions related to functionality, mood, fatigue, sleep, pain, sociability and sexuality. The BETY Scale is a total likert-type scale consisting of 30 items. Each item is scored between 0 and 4, and a high score is associated with poor biopsychosocial status. Responses are rated on a 5-point Likert scale; 4: Always, 3: Often, 2: Sometimes, 1: Rarely, 0: No, never

CONTACTS AND LOCATIONS:
Overall Officials: Aysenur TUNCER, PhD, Study Director — Hasan Kalyoncu University
Locations (1):
- Abdulkadir Konukoğlu Sağlıklı Hayat Merkezi, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No